CLINICAL TRIAL: NCT04812795
Title: Project RESIST: Increasing Resistance to Tobacco Marketing Among Young Adult Sexual Minority Women Using Inoculation Message Approaches
Acronym: RESIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Michigan State University (Other); Harvard School of Public Health (HSPH) (Other); Stanford University (Other); Dana-Farber Cancer Institute (Other); Fenway Community Health (Other)
Responsible Party: Principal Investigator, Andy Tan, Associate Professor, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 843579; R01CA237670 (NIH)
Record Dates: First submitted 2021-03-09; First posted 2021-03-24 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Cigarette Smoking Behavior
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the tailored or non-tailored arms using random assignment function within survey software.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Culturally tailored (Non-smokers) (Experimental): The anti-smoking and anti-industry messages will be culturally tailored to specifically reach out to young adult SMW. They will receive only messages that are culturally tailored at baseline and weeks 1, 2, and 3.
  Culturally tailored anti-smoking messages: Anti-smoking messages that are culturally tailored for sexual minority women.
  Interventions: Other: Culturally tailored anti-smoking messages
- Non-culturally tailored (Non-smokers) (Active Comparator): The anti-smoking and anti-industry messages will not be culturally tailored. They will receive only messages that are not culturally tailored at baseline and weeks 1, 2 and 3.
  Non-culturally tailored interventions: Anti-smoking messages that are not culturally tailored for sexual minority women.
  Interventions: Other: Non-culturally tailored interventions
- Culturally Tailored (Smokers) (Experimental): The anti-smoking and anti-industry messages will be culturally tailored to specifically reach out to young adult SMW. They will receive only messages that are culturally tailored at baseline and weeks 1, 2, and 3.
  Culturally tailored anti-smoking messages: Anti-smoking messages that are culturally tailored for sexual minority women.
  Interventions: Other: Culturally tailored anti-smoking messages
- Non-culturally Tailored (Smokers) (Active Comparator): The anti-smoking and anti-industry messages will not be culturally tailored. They will receive only messages that are not culturally tailored at baseline and weeks 1, 2 and 3.
  Non-culturally tailored interventions: Anti-smoking messages that are not culturally tailored for sexual minority women.
  Interventions: Other: Non-culturally tailored interventions

INTERVENTIONS:
Other: Culturally tailored anti-smoking messages — Anti-smoking messages that are culturally tailored for sexual minority women.
  Arms: Culturally Tailored (Smokers); Culturally tailored (Non-smokers)
Other: Non-culturally tailored interventions — Anti-smoking messages that are not culturally tailored for sexual minority women.
  Arms: Non-culturally Tailored (Smokers); Non-culturally tailored (Non-smokers)

SUMMARY:
Project RESIST is an R01 study funded by NCI focused on determining the effects of using culturally tailored inoculation approaches to increase resilience to tobacco marketing influences among young adult sexual minority women ages 18-30 and incorporates critical stakeholder inputs that support later adoption and implementation. The study team is utilizing formative research to design and pre-test anti-smoking messages and two national longitudinal online survey experiments.

DETAILED DESCRIPTION:
This study will recruit 2000 young adult sexual minority women (SMW), ages 18-30 years, current smokers (n = 1000) and not current smokers (n=1000). The study team will randomly assign participants to a condition in which they will be exposed to either culturally tailored anti-smoking messages or non-tailored. Participants will receive these messages at baseline and 1, 2, and 3 weeks post baseline. They will be asked to complete a follow-up survey one month post baseline. Intentions to quit smoking as well as intention (among current smokers) and intention to purchase cigarettes (among current nonsmokers) will be measured at baseline and one-month post baseline.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-30
* Woman
* Identifies as a sexual minority (any sexual orientation other than heterosexual)
* Lives in the United States
* Able to take surveys in English

Exclusion Criteria:

* Under 18 or older than 30
* Men
* Heterosexual
* Lives outside the United States
* Unable to take survey in English

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Anyone who identifies as a woman, whether they are cisgender or transgender, would meet the gender-based eligibility requirement.
Enrollment: 2214 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-06-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Zulkiewicz BA, Chen JT, Hanby EP, Ramanadhan S, Obedin-Maliver J, Lunn MR, Scout NFN, Gordon B, Applegate J, Machado A, Viswanath K, Potter J, Liu S, Tan ASL. Anti-industry beliefs and attitudes mediate the effect of culturally tailored anti-smoking messages on quit intentions among sexual minority women. Sci Rep. 2024 Nov 15;14(1):28084. doi: 10.1038/s41598-024-78207-7. PMID 39543185
- [Derived] Tan ASL, Chen JT, Keen R, Scout N, Gordon B, Applegate J, Machado A, Hanby E, Liu S, Zulkiewicz B, Ramanadhan S, Obedin-Maliver J, Lunn MR, Viswanath K, Potter J. Culturally Tailored Anti-Smoking Messages: A Randomized Trial With U.S. Sexual Minority Young Women. Am J Prev Med. 2024 May;66(5):840-849. doi: 10.1016/j.amepre.2023.12.001. Epub 2023 Dec 7. PMID 38065403

RESULTS

PARTICIPANT FLOW:
Groups:
- Culturally Tailored (Non-smokers); Culturally Tailored (Smokers): The anti-smoking and anti-industry messages will be culturally tailored to specifically reach out to young adult sexual minority women. They will receive only messages that are culturally tailored at baseline and weeks 1, 2, and 3.
  Culturally tailored anti-smoking messages: Anti-smoking messages that are culturally tailored for sexual minority women.
Period: Overall Study
Arm/Group | Culturally Tailored (Non-smokers) | Non-culturally Tailored (Non-smokers) | Culturally Tailored (Smokers) | Non-culturally Tailored (Smokers)
Started | 501 | 501 | 613 | 599
Completed | 407 | 401 | 492 | 476
Not Completed | 94 | 100 | 121 | 123

BASELINE CHARACTERISTICS:
Population: U.S. young adult sexual minority women ages 18-30.
Groups:
- Total: Total of all reporting groups
Arm/Group | Culturally Tailored (Non-smokers) | Non-culturally Tailored (Non-smokers) | Culturally Tailored (Smokers) | Non-culturally Tailored (Smokers) | Total
Number analyzed (Participants) | 501 | 501 | 613 | 599 | 2214
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.90 (3.47) | 23.7 (3.73) | 24.82 (2.91) | 24.77 (2.90) | 24.33 (3.27)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 15 | 13 | 26 | 17 | 71
  Female | 486 | 488 | 587 | 578 | 2139
  Unknown | 0 | 0 | 0 | 4 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 74 | 73 | 57 | 58 | 262
  Not Hispanic or Latino | 427 | 428 | 556 | 541 | 1952
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 90 | 69 | 167
  Asian | 38 | 43 | 45 | 44 | 170
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 2 | 3
  Black or African American | 34 | 32 | 80 | 77 | 223
  White | 356 | 362 | 381 | 380 | 1479
  More than one race | 66 | 52 | 16 | 24 | 158
  Unknown or Not Reported | 3 | 8 | 0 | 3 | 14
Intention to quit smoking [Mean (Standard Deviation); unit: units on a scale] — We used a 4-item scale on intention to quit smoking at baseline and at one-month follow-up among current smokers only: 1) I will make an effort to quit smoking in the next 30 days; 2) I intend to quit smoking in the next 30 days; 3) I expect to quit smoking in the next 30 days; 4) How likely is it that you will quit smoking in the next 30 days.
  Responses ranged on 7-point Likert-like scales.
  Responses were summed to create a scale for intention to quit (range from 4-28).
  Higher values indicate greater intention to quit smoking in the next 30 days. Population: Non-smokers were not asked the questions about intentions to quit smoking.
  units on a scale
    number analyzed (Participants) | 0 | 0 | 613 | 599 | 1212
    (all) |  |  | 16.54 (5.83) | 16.35 (5.87) | 16.44 (5.85)
Intention to purchase cigarettes [Mean (Standard Deviation); unit: units on a scale] — We used the Juster scale to measure intention to purchase cigarettes at baseline and at one-month follow-up.
  Participants were asked, "How likely are you to purchase cigarettes in the next 6 months?"
  Responses ranged from 0=No chance, almost no chance (1 in 100) to 10=Certain, practically certain (99 in 100).
  Higher values reflect higher intention to purchase.
  units on a scale | 0.47 (1.37) | 0.39 (1.18) | 7.42 (2.59) | 7.36 (2.59) | 4.24 (4.05)

OUTCOME MEASURES:

1. Primary Outcome: Intention to Quit Smoking
Description: Intention to quit smoking will be measured using the Burkhalter intention to quit smoking four item scale that measures readiness to cut down or quit smoking in the next 30 days at baseline and 1 month follow-up.
  Participants were asked to rate 4 statements: I will make an effort to quit smoking in the next 30 days (Unlikely to Likely); I intend to quit smoking in the next 30 days (Strongly disagree to Strongly Agree); I expect to quit smoking in the next 30 days (Definitely false to Definitely true); How likely is it that you will quit smoking in the next 30 days (Unlikely to Likely). Responses ranged on 7-point Likert-like scales. Responses were summed to create a scale for intention to quit (range from 4-28).
  This will only be measured among current smokers. Lowest score is 4 and highest mean score is 28. Higher scores indicate increased intention to quit smoking within the next 30 days.
Time Frame: Day 30
Population: U.S. young adult sexual minority women who smoked at least one cigarette in the past 30 days as baseline.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Culturally Tailored (Non-smokers) | Non-culturally Tailored (Non-smokers) | Culturally Tailored (Smokers) | Non-culturally Tailored (Smokers)
Number analyzed (Participants) | 0 | 0 | 489 | 469
Score on a scale |  |  | 4.814 (5.199) | 4.844 (4.966)

2. Primary Outcome: Change in Intention to Purchase Cigarettes
Description: The Juster scale was used to measure intention to purchase cigarettes at baseline and at one-month follow-up.
  Participants were asked, "How likely are you to purchase cigarettes in the next 6 months?" Responses ranged from 0=No chance, almost no chance (1 in 100) to 10=Certain, practically certain (99 in 100).
  Higher values reflect higher intention to purchase.
Time Frame: Day 30
Population: U.S. young adult sexual minority women who completed the follow-up survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Culturally Tailored (Non-smokers) | Non-culturally Tailored (Non-smokers) | Culturally Tailored (Smokers) | Non-culturally Tailored (Smokers)
Number analyzed (Participants) | 407 | 401 | 492 | 476
units on a scale | -0.034 (1.261) | -0.110 (1.050) | -2.195 (2.954) | -2.313 (2.837)

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- Culturally Tailored (Current Smokers): The anti-smoking and anti-industry messages will be culturally tailored to specifically reach out to young adult SMW. They will receive only messages that are culturally tailored at baseline and weeks 1, 2, and 3.
  Culturally tailored anti-smoking messages: Anti-smoking messages that are culturally tailored for sexual minority women.
- Non-culturally Tailored (Current Smokers): The anti-smoking and anti-industry messages will not be culturally tailored. They will receive only messages that are not culturally tailored at baseline and weeks 1, 2 and 3.
  Non-culturally tailored interventions: Anti-smoking messages that are not culturally tailored for sexual minority women.
Arm/Group | Culturally Tailored (Non-smokers) | Non-culturally Tailored (Non-smokers) | Culturally Tailored (Current Smokers) | Non-culturally Tailored (Current Smokers)
All-Cause Mortality (participants affected / at risk) | 0/501 | 0/501 | 0/613 | 0/599
Serious Adverse Events (participants affected / at risk) | 0/501 | 0/501 | 0/613 | 0/599
Other Adverse Events (participants affected / at risk) | 0/501 | 0/501 | 0/613 | 0/599

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-17): https://cdn.clinicaltrials.gov/large-docs/95/NCT04812795/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT04812795/ICF_001.pdf